CLINICAL TRIAL: NCT01918202
Title: A Phase 1, Open-label Adaptive Design Study To Evaluate Pde10 Enzyme Occupancy As Measured By Positron Emission Tomography (Pet) Following Single Oral Dose Administration Of Pf-02545920 In Healthy Male Subjects
Brief Title: A Study To Evaluate The PDE10 Enzyme Occupancy Following A Single Dose Of PF-02545920 In Healthy Male Volunteers
Acronym: PET
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: A8241017; 2013-002733-38 (EudraCT Number)
Record Dates: First submitted 2013-08-05; First posted 2013-08-07 (Estimated); Last update posted 2014-11-10 (Estimated); Status verified 2014-11

CONDITIONS: Healthy
Keywords: Enzyme occupancy; PET; Phosphodiesterase 10 inhibitor
MeSH Terms: interventions — 2-((4-(1-methyl-4-pyridin-4-yl-1H-pyrazol-3-yl)phenoxy)methyl)quinoline

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Cohort 1 - 20 mg (Experimental): Cohort will include 4 HVs/completers who will receive a single 20 mg dose of PF-02545920.
  Interventions: Drug: 20 mg PF-02545920
- Cohort 2 ( adaptive dose, optional) (Experimental): Cohort 2 will include 4 HVs/completers who will receive a single dose of PF-02545920. The dose will be selected based on the results obtained for Cohort 1.
  Interventions: Drug: PF-02545920
- Cohort 3 ( adaptive dose, optional) (Experimental): Cohort 3 will include 4 HVs/completers who will receive a single dose of PF-02545920. The dose will be selected based on the results obtained for Cohort 1.
  Dose options range from 30 mg to 10 mg, 5 mg, 2mg, 1 mg. This cohort is optional
  Interventions: Drug: PF-02545920

INTERVENTIONS:
Drug: 20 mg PF-02545920 — Subject will receive a single dose of 20 mg PF-02545920.
  Arms: Cohort 1 - 20 mg
Drug: PF-02545920 — The dose will be selected based on the results obtained for Cohort 1. Dose options range from 30 mg to 10 mg, 5 mg, 2mg, 1 mg.
  This cohort is optional.
  Arms: Cohort 2 ( adaptive dose, optional)
Drug: PF-02545920 — The dose will be selected based on the results obtained for Cohort 1 and cohort 2.
  Arms: Cohort 3 ( adaptive dose, optional)

SUMMARY:
This Phase 1 study will evaluate PDE10 enzyme occupancy using Positron Emission Tomography after a single dose of PF-02545920 in Healthy male volunteers.

ELIGIBILITY:
Inclusion Criteria:

* healthy male volunteers

Exclusion Criteria:

* History of orthostatic hypotension
* History of prior radiation exposure for research purposes, or radiation therapy

Ages: 21 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2014-03; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Central PDE10A enzyme occupancy values in the striatum. | Day 10
  Using Positron Emission Tomography and a radiotracer (MNI-659) for PF-02545920, the central PDE10A enzyme occupancy values will be measured in the striatum at different single oral doses of PF-02545920.

SECONDARY OUTCOMES:
Central PDE10A enzyme occupancy values in the globus pallidus, in the caudate and in the putamen (separately). | Day 10
  Using Positron Emission Tomography and a radiotracer (MNI-659) for PF-02545920, central PDE10A enzyme occupancy values in the globus pallidus, in the caudate and in the putamen be measured (separately) at different single oral doses of PF-02545920.
Maximum Observed Plasma Concentration (Cmax) | Day 10
  Cmax for serum PF-02545920 during the post-dose positron emission tomography (PET) scan.
Time to Reach Maximum Observed Plasma Concentration (Tmax) | Day 10
  Tmax for serum PF-02545920 during the post-dose positron emission tomography (PET) scan.
Average serum concentration | Day 10
  Average serum 02545920 during the post-dose positron emission tomography (PET) scan.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Karolinska Trial Alliance (KTA) M62, Huddinge, Stockholm County, Sweden

REFERENCES:
- [Derived] Delnomdedieu M, Forsberg A, Ogden A, Fazio P, Yu CR, Stenkrona P, Duvvuri S, David W, Al-Tawil N, Vitolo OV, Amini N, Nag S, Halldin C, Varrone A. In vivo measurement of PDE10A enzyme occupancy by positron emission tomography (PET) following single oral dose administration of PF-02545920 in healthy male subjects. Neuropharmacology. 2017 May 1;117:171-181. doi: 10.1016/j.neuropharm.2017.01.016. Epub 2017 Jan 22. PMID 28122201
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A8241017&StudyName=A%20Study%20To%20Evaluate%20The%20PDE10%20Enzyme%20Occupancy%20Following%20A%20Single%20Dose%20Of%20PF-02545920%20In%20Healthy%20Male%20Volunteers